CLINICAL TRIAL: NCT04978857
Title: Feasibility Study of Virtual Reality to Promote the Awakening of Patients in a State of Minimal Consciousness
Acronym: REVEIL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 49RC20_0238
Record Dates: First submitted 2021-07-23; First posted 2021-07-27 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Consciousness Disorder
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual reality headset (Experimental)
  Interventions: Other: autobiographic movie

INTERVENTIONS:
Other: autobiographic movie — viewing an autobiographic film through a virtual reality headset

SUMMARY:
Advances in neurosurgery and neuroresuscitation have improved patients' prognosis. However, 2% of serious head injuries progress to a vegetative state, this condition persisting at 1 year for 1% of these patients.

The minimum state of consciousness is to be distinguished from coma and vegetative state, it is a condition marked by a severe alteration of consciousness in which there are minimal and fluctuating, but obvious, signs of environmental consciousness. There is a minimum degree of response to some stimulations, response generally fluctuating over time. In practice, these patients are unable to consistently follow simple instructions, but they often have a preserved visual pursuit (proper rotation of the head when someone enters the room, prolonged eye follow-up, etc.). Patients with minimal awareness have been shown to perceive emotions and pain. These patients may exhibit behavioural and emotional changes (smiling, crying motivated), induced by verbal stimulations (familiar voice). But these events remain fluctuating during the day or according to the days and interlocutors.

For the moment, the most commonly accepted strategy since the 1990s remains sensory stimulation (SS), while knowing that this term includes extremely varied stimulations (sensory, olfactory, auditory, fixation on a mirror, etc.) without the practice of this technique being well defined and systematized.

It has been shown that a regular family visit program with auditory, emotional and tactile stimuli improves the state of consciousness of these patients. Physicians also know that this SS must be personalized and adapted to the patient's tolerance and premorbid preferences.

SS programmes are poorly standardized. Programmes generally consist of a simple, moderate to high intensity, non-standardized stimulation, presented repetitively and frequently. Indeed, it has been shown that stimulation must begin early, be frequent, and continue until reactions appear.

In this project, investigator want to use the new technologies now commonly used such as photos, videos or sounds taken by smartphone's relatives of the brain patient-injured in order to make a personalized 3D film using film editing software and a predefined film frame, by integrating autobiographical elements and emotional, multisensory (binaural sound, vibration) integrating, if possible, a certain interactivity (haptic feedback, triggering of videos by the patient's eyes).

The objective is to develop an innovative multi-sensory stimulation technique through a personalised enriched environment to induce, facilitate and accelerate the return to consciousness of patients in altered state of consciousness during their initial management.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with minimal consciousness
* Patient affiliated or beneficiary of a social security scheme
* Signature of consent by a relative of the patient
* Tolerance of the multisensory stimulation material during the pre-inclusion phase

Exclusion Criteria:

* Minor
* Pregnant woman
* Patient with contraindication to study procedures (Contraindication to wearing a virtual reality headset (unbalanced epilepsy, craniofacial trauma, major visual disturbances; contraindication to the fMRI)
* Person deprived of liberty by judicial or administrative decision
* Person receiving psychiatric care under duress

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2025-11-13 (Estimated); Study Completion 2026-03-13 (Estimated)

PRIMARY OUTCOMES:
percentage of patients without any adverse event or sign of bad tolerance | 1 month
  to assess the feasibility of multisensory virtual reality stimulation proposed in this study in patients with minimal post-traumatic consciousness

SECONDARY OUTCOMES:
Time required for film design | 2 weeks
  to assess the feasibility of making a personalized film
type and quantity of autobiographical material to be obtained from the patient's relatives | 2 weeks
  to assess the feasibility of making a personalized film
Patient clinical responses (blood pressure, body motion, eye-tracking) | 1 month
  To assess signs of patient's interaction with the virtual reality headset during the pre-inclusion phase and during the test phase, and the evolution over time of these signs during the test phase
Wessex Head Injury Matrix (WHIM) | 6 month
  To assess the evolution of the patient's clinical status Scale from 0 which means vegetative state to 62 which means pauci-relational state
Coma Recovery Scale - Revised (CRS-R) | 6 month
  To assess the evolution of the patient's clinical status
functional MRI | 1 month
  To assess and compare the different brain networks identified during the fMRI performed one week after the initial fMRI test phase performed the week preceding the test phase.
patient's relative satisfaction scale | 1 month
  To assess patient's family's feelings and experiences with this intervention (interviews etc).
  Scale from 1 (minimum) to 7 (maximum); 1 means not satisfied at all and 7 means very satisfied
healthcare team satisfaction scale | 1 month
  To assess healthcare team feelings and experiences with this intervention (adherence to this rehabilitation technique etc) Scale from 1 (minimum) to 7 (maximum); 1 means not satisfied at all and 7 means very satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Angers, Angers, France